**Official Title:** A Prospective, Randomized, Double-masked, Active Comparator controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared with Intravitreal Aflibercept in Participants with Neovascular (Wet) Age-related Macular Degeneration (wAMD)

NCT Number: NCT04964089

**Document Date:** SAP Version 1.0, 20 June 2023

# STATISTICAL ANALYSIS PLAN

A Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared with Intravitreal Aflibercept in Participants with Neovascular (Wet) Agerelated Macular Degeneration (wAMD) (DAYLIGHT)

| Sponsor: | Kodiak Sciences Inc.<br>1200 Page Mill Road<br>Palo Alto, CA 94304 USA |
|---|---|
| Sponsor Contact<br>& Medical Monitor: | Kodiak Sciences Inc. |
| IND Number: | 136167 |
| Protocol Numbers: | KS301P107 |
| EUDRACT Number: | 2021-000225-27 |
| Test Product: | KSI-301 (tarcocimab tedromer) |
| Statistical Analysis Plan Version: | 1.0 |
| Statistical Analysis Plan Version Date: | June 20, 2023 |
| Supersedes: | N/A |

#### **CONFIDENTIAL**

The information in this document is confidential and may not be disclosed to others in whole or in part without express, written authorization from Kodiak Sciences Inc., except to the extent necessary to obtain informed consent from persons receiving the investigational drug or their legal guardians, or for discussions with local regulatory authorities, institutional review boards (IRB) or persons participating in the conduct of the trial.

# **SPONSOR SIGNATORY**

| Study Title: | A Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared with Intravitreal Aflibercept in Participants with Neovascular (Wet) Age-related Macular Degeneration (wAMD) (DAYLIGHT) |
|---|---|
| Protocol Code: | KS301P107 |
| Statistical Analysis Plan Version: | 1.0 |
| Statistical Analysis Plan Version Date: | June 20, 2023 |
| Prepared by: | |

| Statistical Analysis Plan Accepted and Approved by: | |
|---|---|
| Kodiak Sciences Inc.<br>1200 Page Mill Rd.<br>Palo Alto, CA 94304 | Date |
| Kodiak Sciences Inc.<br>1200 Page Mill Rd.<br>Palo Alto, CA 94304 | Date |

# **TABLE OF CONTENTS**

| <b>STA</b> | TISTIC | CAL ANA | ALYSIS PLAN | 1 |
|---|---|---|---|---|
| SPO | NSOR | SIGNAT | ORY | 2 |
| TAB | LE OF | CONTE | NTS | 3 |
| LIST | OF T | ABLES | | 4 |
| LIST | OF A | BBREVIA | ATIONS | 6 |
| 1.0 | INT | RODUCT | TION | 8 |
| 2.0 | STU | DY OBJE | ECTIVES AND ENDPOINTS | 8 |
| 3.0 | INV | <b>ESTIGAT</b> | ΓΙΟΝAL PLAN | 9 |
| | 3.1 | Study I | Design | 9 |
| | 3.2 | Study In | nterventions | 10 |
| | 3.3 | | nization and Stratification | |
| 4.0 | TYP | | LANNED ANALYSES | |
| | 4.1 | | Ionitoring Committee Analyses | |
| | 4.2 | | Analyses | |
| | 4.3 | | nalysis | |
| <b>5.0</b> | GEN | | TATISTICAL METHODS | |
| | 5.1 | - | ing Conventions | |
| | 5.2 | | rd Calculations | |
| | 5.3 | | Definitions and Derived Variables | |
| | 5.4 | • | is Sets | |
| | | 5.4.1 | 3 | |
| | | 5.4.2 | Safety Analysis Set | |
| | 5.5 | | nation of Subgroups | |
| | 5.6 | | le Comparisons/Multiplicity | |
| | 5.7 | | enter Study | |
| | 5.8 | • | is Visit | |
| 6.0 | BAS | | NALYSES | |
| | 6.1 | - | ition of Subjects | |
| | 6.2 | _ | raphic and Other Baseline Characteristics | |
| | | 6.2.1 | Demographics and Baseline Characteristics | |
| | | 6.2.2 | Ocular and Other Medical History | |
| | | 6.2.3 | Prior and Concomitant Medications/Procedures | 17 |

| | 6.3 | Protocol Deviations | 19 |
|---|---|---|---|
| 7.0 | EFFI | CACY ANALYSES | 19 |
| | 7.1 | Primary Efficacy Analysis | |
| | | 7.1.1 Primary Estimand | 19 |
| | | 7.1.2 Analysis of Primary Efficacy Endpoint | 21 |
| | | 7.1.3 Sensitivity Analysis 1 | 21 |
| | | 7.1.4 Sensitivity Analysis 2 (Trimmed Mean Analysis) | 21 |
| | | 7.1.5 Sensitivity Analysis 3 (Tipping Point Analysis) | 23 |
| | 7.2 | Secondary Efficacy Analyses | 24 |
| | | 7.2.1 Analysis of Binary Data | 24 |
| | 7.3 | Exploratory Analyses | 26 |
| | 7.4 | Subgroup Analyses | 27 |
| 8.0 | SAFI | ETY EVALUATION | 27 |
| | 8.1 | Exposure to Study Medication | 27 |
| | 8.2 | Adverse Events | 27 |
| | 8.3 | Deaths, Serious Adverse Events, and other Significant Adverse Events | 29 |
| | 8.4 | Pregnancies | 29 |
| | 8.5 | Intraocular Pressure | 29 |
| | 8.6 | Clinical Laboratory Evaluations | 29 |
| | 8.7 | Vital Signs. | 29 |
| 9.0 | SAM | PLE SIZE CONSIDERATIONS | 30 |
| 10.0 | | MARY OF CHANGES IN THE CONDUCT OF THE STUDY OR | |
| | | NNED ANALYSES | |
| 11.0 | | ERENCES | |
| 12.0 | | ENDICES | |
| | Appe | ndix 1: Schedule of Activities | 32 |

# LIST OF TABLES

| Table 1: Objectives ar | d Endpoints |
|------------------------|-------------|
| Table 2: Subgroups | 14 |

| KS301P107 | SAP | Version | 1.0 |
|---------------|-------|-----------|-----|
| XSI_301 - Kod | iak S | ciences l | ne |

## CONFIDENTIAL

| Table 3: Windows for Unscheduled Visit | .15 |
|--------------------------------------------------------------|-----|
| Table 4: Secondary Efficacy Endpoints and Analysis Methods | .25 |
| Table 5: Exploratory Efficacy Endpoints and Analysis Methods | .26 |

# LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|--------------------------------------------------|
| ANCOVA | Analysis of covariance |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| AI | Artificial intelligence |
| ALT | Alanine aminotransferase |
| AMD | Age-related Macular Degeneration |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| ATE | Arteriothromboembolic |
| BCVA | Best-corrected visual acuity |
| BP | Blood pressure |
| CI | Confidence Interval |
| CMH | Cochran-Mantel-Haenszel |
| CNV | Choroidal Neovascularization |
| CSR | Clinical Study Report |
| CST | Central Subfield Thickness |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| ET | Early Termination |
| ETDRS | Early treatment diabetic retinopathy study |
| FA | Fluorescein angiography |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| FP | Fundus photography |
| ICE | Intercurrent event |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IND | Investigational New Drug (application) |
| IOI | Intraocular inflammation |
| IOP | Intraocular Pressure |
| IRB | Institutional Review Board |
| IRT | Interactive Response Technology |
| ITP | Individualized Treatment Period |
| LOQ | Level of Quantification |
| MAR | Missing at Random |
| MNAR | Missing not at Random |
| MedDRA | The Medical Dictionary for Regulatory Activities |
| MMRM | Mixed Model for Repeated Measures |
| NI | Non-Inferiority |

| Abbreviation | Definition |
|--------------|------------------------------------|
| OCT | Optical Coherence Tomography |
| PT | Preferred Term |
| RAP | Retinal Angiomatous Proliferations |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SOC | System Organ Class |
| TEAE | Treatment Emergent AE |
| ULN | Upper Limits of Normal |
| VA | Visual acuity |
| VEGF | Vascular Endothelial Growth Factor |
| VRC | Vienna Reading Center |
| WHO | World Health Organization |

#### 1.0 INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide a comprehensive and detailed description of the methods and presentation of data analyses for Study KS301P107 (Protocol Amendment 2.0, dated 16 March 2022), A Prospective, Randomized, Double-masked, Active Comparator-controlled, Multi-center, Two-arm, Phase 3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 Compared with Intravitreal Aflibercept in Participants with Neovascular (Wet) Age-related Macular Degeneration (wAMD) (DAYLIGHT). This study is conducted in accordance with the protocols, Good Clinical Practice, the Declaration of Helsinki, and any other applicable regulatory requirements.

Descriptions of planned analyses are provided *a priori* to preserve the validity of the interpretation of the statistical analysis results pertaining to the primary and secondary efficacy endpoints. The statistical methods applied in the design and planned analyses are consistent with the International Council for Harmonisation (ICH) guidelines *Statistical Principles for Clinical Trials* (E9) (1998) and ICH E9 (R1) *Addendum on Estimands and Sensitivity Analysis in Clinical Trials to the Guideline on Statistical Principles for Clinical Trials* (2020).

This SAP provides details of the statistical analysis results to be presented in the clinical study reports (CSR). Analyses of pharmacokinetics, biomarkers, and anti-drug antibodies will be addressed in separate analysis plan(s).

Any changes between the statistical methods and study endpoints provided in the clinical study protocol and this SAP will be described and explained in Section 10.0; any changes or deviations from this SAP relative to the final analyses will be fully documented in the CSR. Minor changes or deviations from the templates for tables, figures, and listings need not be documented in the CSR.

#### 2.0 STUDY OBJECTIVES AND ENDPOINTS

Table 1 lists the primary and secondary study objectives, along with their corresponding endpoints.

Table 1: Objectives and Endpoints

| Objectives | Corresponding Endpoints |
|---|---|
| Primary | |
| To demonstrate that KSI-301 5 mg is non-inferior to aflibercept 2 mg, with respect to the change in best corrected visual acuity (BCVA) from Day 1 to the average of Weeks 40, 44, and 48. | Mean change in BCVA from baseline (Day 1) to the<br>average of Weeks 40, 44, and 48, in Early Treatment<br>Diabetic Retinopathy Study (ETDRS) Letters. |
| Secondary | |
| To evaluate the efficacy of KSI-301 5 mg compared to aflibercept 2 mg over the study duration by assessing visual parameters. | Mean change in BCVA (ETDRS Letters) from baseline (Day 1) by visit over time. |
| | <ul> <li>Proportion of participants who gain ≥5, ≥10 and ≥15<br/>letters from baseline (Day 1) by visit over time.</li> </ul> |
| | <ul> <li>Proportion of participants who lose ≥5, ≥10 and ≥15<br/>letters from baseline (Day 1) by visit over time.</li> </ul> |
| | <ul> <li>Proportion of participants with BCVA Snellen<br/>equivalent of 20/40 or better from baseline (Day 1) over<br/>time.</li> </ul> |
| | <ul> <li>Proportion of participants with BCVA Snellen<br/>equivalent of 20/200 or worse from baseline (Day 1)<br/>over time.</li> </ul> |
| To evaluate the efficacy of KSI-301 5 mg compared to aflibercept 2 mg over the study duration by assessing anatomical parameters. | Mean change in optical coherence tomography (OCT) central subfield thickness (CST) and other morphological parameters from baseline (Day 1) to the average of Weeks 40, 44, and 48 and over time. |
| To evaluate the safety and tolerability of KSI-301 5 mg compared to aflibercept 2 mg. | Incidence of ocular and systemic adverse events up to<br>Week 52. |

#### 3.0 INVESTIGATIONAL PLAN

## 3.1 Study Design

This is a Phase 3, prospective, randomized, double-masked, two-arm, multi-center study evaluating the efficacy and safety of repeated intravitreal dosing of KSI-301 5 mg in patients with treatment naïve wAMD. A brief description of the study design and study treatment regimen appears below; additional details can be found in the study protocol.

The schedule of activities is provided in Appendix 1.

The overall duration of the study is approximately 52 weeks after the last participant is randomized to the study. Participant duration is defined as the date a signed written informed consent is provided through the last safety follow-up visit at Week 52. Thus, participant duration is approximately 55 weeks and includes a screening period of up to 21 days (Days -21 to -1), a treatment period of approximately 44 weeks (Day 1 to Week 44), a 4-week follow-up period for

safety and efficacy assessments at Week 48, and a final follow-up for safety assessments at Week 52

The primary endpoint is defined as the mean change in ETDRS BCVA from baseline (Day 1) to the average of Weeks 40, 44, and 48.

A single eye per participant will be designated as the Study Eye. If both eyes are eligible to become the Study Eye, the eye with worse BCVA at Screening will be selected as the Study Eye. If both eyes are eligible and have the same BCVA, the decision of which eye to select as the Study Eye will be made by the Investigator.

Participants will be randomly assigned (1:1) into one of two treatment groups:

- o KSI-301 5 mg, or
- o Aflibercept 2 mg.

## 3.2 Study Interventions

Study interventions are summarized in the Protocol Table 2.

#### 3.3 Randomization and Stratification

Patients who meet all inclusion criteria and none of the exclusion criteria will be centrally assigned to a randomized study intervention using an Interactive Response Technology (IRT) system. Randomization will be stratified by

#### 4.0 TYPES OF PLANNED ANALYSES

#### 4.1 Data Monitoring Committee Analyses

An Independent Data Monitoring Committee (IDMC) will monitor study conduct and safety on an ongoing basis. Members of the IDMC will be external to the Sponsor and will follow a charter that outlines the IDMC membership and responsibilities, the timing of IDMC meetings, the content of the analysis report for the IDMC meetings, and the communication with the Sponsor. The IDMC can recommend changes to the conduct of the study based on the evaluated data and may recommend stopping the study early for safety reasons only as detailed in the charter.

## 4.2 Interim Analyses

No interim analyses were planned or performed.

## 4.3 Final Analysis

The final analysis will be performed when all patients have either completed all phases of the study or have discontinued the study prematurely.

#### 5.0 GENERAL STATISTICAL METHODS

SAS (SAS Institute Inc., Cary NC, USA) Version 9.4 or higher will be used for the study analyses.

# 5.1 Reporting Conventions

Tables and figures will be summarized by treatment group. Tables summarizing demographics and other baseline characteristics will also include a column for all patients combined. In general, all data collected and any derived data will be presented in subject data listings, for all randomized patients. Listings will be ordered by treatment group, subject number, and assessment or event date. The treatment groups will be displayed in the same order as the summary tables. The treatment groups presented in listings will be based on the planned assignment, unless otherwise noted.

In general, continuous variables will be summarized to indicate the study population sample size (N), number of subjects with available data (n), mean, SD, median, 25th (Q1) and 75th (Q3) quartiles, minimum, and maximum values. Categorical variables will be summarized by the population size (N), number of subjects with available data (n), number of subjects in each category, and the percentage of subjects in each category. Unless otherwise noted, the denominator to determine the percentage of subjects in each category will be based on the number of subjects with available data. The denominator for percentages for incidence data (such as adverse events) will be based on the number of subjects in the analysis population "at risk." Select ordinal data may be summarized using both descriptive statistics and counts and percentages of subjects in each category, as appropriate.

Non-zero percentages will be rounded to one decimal place. Percentages that round down to 0 or up to 100% will be displayed as "<0.1%" and ">99.9%", respectively. Rounding conventions for presentation of summary statistics will be based on the precision of the variable of summarization, as it is collected in its rawest form e.g., on the electronic case report form (eCRF) and are outlined as follows:

- The mean and median will be rounded to an additional decimal place than the precision of the variable of summarization;
- Measures of variability (e.g., SD, SE) will be rounded to two additional decimal places than the precision of the variable of summarization; and
- o Minimum and maximum values will be presented using the same precision as the variable of summarization.

Other statistics (e.g., CIs) will be presented using the same general rules outlined above or assessed for the most appropriate presentation based on the underlying data.

Unless noted otherwise, statistical significance testing will be two-sided and performed using  $\alpha$ =0.05. Confidence intervals (CIs) will be calculated at the 95% level, reflecting a type I error rate of 0.05. P-values will be reported for all statistical tests, rounded to four decimal places. P-values less than 0.0001 will be displayed as "<0.0001"; p-values greater than 0.9999 will be displayed as ">0.9999".

#### 5.2 Standard Calculations

Where appropriate, the calculated study day will be presented with the assessment or event date on subject data listings. Study day will be determined as:

- The assessment/event date minus the date of first dose of study drug, if the assessment/event date is prior to the date of first dose; and
- o The assessment/event date minus the date of first dose of study drug, plus one, if the assessment/event date is on or after the date of first dose.

Start and stop dates will be imputed when partial dates are present as needed, to determine treatment emergent events and concomitant medications/procedures. No imputations will be done for a completely missing start/stop date or for subjects who did not receive study treatment.

Start dates with a missing day but with month and year available will be imputed such that:

- o If the provided month and year match the month and year for that subject's first dose date, then the Day 1 date will be used.
- o In all other cases the 1st of the month will be used with the provided month and year.

Start dates with a missing day and month but with available year will be imputed such that:

- o If the provided year matches the year for that subject's first dose date, then the first dose date will be used.
- o In all other cases the 1st of January will be used with the provided year.

Stop dates will be imputed as follows:

- o Missing day with a provided year and month will use the last day of the month.
- o Missing day and month with provided year will use December 31.

If the imputed stop date is greater than the last study date for the subject, then the imputed date will be replaced with the last available event date for the subject in the study.

Other variables requiring calculations will be derived using the following formulas:

- O Days: A duration between two dates expressed in days will be calculated using the following conventions:
  - Later date earlier date + 1.
- o Months: A duration expressed in months will be calculated by dividing the duration in days by (365.25 /12).
- Years: A duration expressed in years will be calculated by dividing the duration in days by 365.25.

## 5.3 Study Definitions and Derived Variables

Baseline values are defined as the most recent values prior to the first dose of study treatment.

#### 5.4 Analysis Sets

The efficacy and safety analyses that are specified in Sections 7.0 and 8.0 will utilize the analysis sets as specified in this section.

#### 5.4.1 Full Analysis Set

The Full Analysis Set (FAS) includes all patients who received any study treatment (KSI-301 or aflibercept). Patients will be analyzed according to their randomized treatment. The FAS will be used in the primary analysis of efficacy.

#### 5.4.2 Safety Analysis Set

The Safety Analysis Set includes all patients who received any study treatment (KSI-301 or aflibercept). Patients will be analyzed according to the study treatment they actually received.

#### 5.5 Examination of Subgroups

The primary efficacy endpoints will be summarized in the following subgroups of baseline characteristics.

**Table 2: Subgroups** 

| Characteristics | Subgroup |
|----------------------|-------------------------------------------|
| Age | 10.64 |
| | • 18-64 years of age |
| | 65-74 years of age |
| | 75-84 years of age |
| | • ≥85 years of age |
| | • < 65 years of age |
| | • ≥ 65 years of age |
| | <ul> <li>&lt; 75 years of age</li> </ul> |
| | • ≥ 75 years of age |
| Sex | • Female |
| | • Male |
| Ethnicity | Hispanic or Latino |
| | Not Hispanic or Latino |
| BCVA* | BCVA: 83-70 letters |
| | BCVA: 69-50 letters |
| | • BCVA: ≤ 49 letters |
| Geographic location* | North America |
| | Rest of World |
| Race | White |
| | Black or African American |
| | Asian |
| | American Indian or Alaska Native |
| | Native Hawaiian or other Pacific Islander |
| - | Other |
| Lens status | Phakic |
| | Pseudophakic |
| | Aphakic |
| | • |

| Characteristics | Subgroup |
|-----------------|----------|

Other subgroup analyses may be explored as needed.

## 5.6 Multiple Comparisons/Multiplicity

#### 5.7 Multicenter Study

This is a multicenter, international study. Efficacy data collected from all study sites will be pooled for data analysis. The effect of study site on the efficacy analysis results may be explored, as needed.

#### 5.8 Analysis Visit

For efficacy analyses, unscheduled or early termination visits will be assigned a study day and then mapped to the appropriate analysis window as detailed in Table 3. In the event where more than one record falls in the same analysis window, the following rules will be used in sequential order to determine the record that will be used for data analysis:

- If there is a scheduled visit in the analysis window, then the scheduled visit's data will be used.
- If there is no scheduled visit in the analysis visit window, the record that is the closest to the scheduled study day at a given visit will be used.
- If there is no scheduled visit in the analysis visit window and there is a tie between the two records with regards to the number of days before and after the scheduled study day, the later record will be used.

Analysis visit windows will not apply to subject data listings. Prior to any missing data imputations or analysis, the analysis visit windows will be applied to the data.

Table 3: Windows for Unscheduled Visit

| | Scheduled | Starting Day for | Ending Day for |
|------------------|-----------|------------------|----------------|
| Nominal Visit | Study Day | Nominal Visit | Nominal Visit |
| Day 1 | 1 | 1 | 1 |
| Week 2 | 14 | 2 | 21 |
| Week 4 | 28 | 22 | 42 |
| Week 8 – Week 52 | Week×7 | (Week×7)-13 | (Week×7)+14 |

Note: Nominal visits are at Day 1, Weeks 2, 4, 8, ... every 4 weeks from Week 8 until Week 52.

#### 6.0 BASELINE ANALYSES

## 6.1 Disposition of Subjects

Subject disposition will be summarized by treatment group and overall. The following will be summarized:

- The number of patients screened
- The number of patients randomized
- The number of patients (%) in the Full Analysis Set
- The number of patients (%) in the Safety Analysis Set
- The number of patients (%) completing study treatment
- The number of patients (%) discontinuing the study treatment and the reasons for discontinuation of study treatment
- The number of patients (%) discontinuing study and the reasons for discontinuation of study

Subject disposition will also be summarized separately for each study site. Subject completion status, date of study completion/discontinuation, study day of discontinuation, and reason for discontinuation will be listed.

Patients who did not meet inclusion or exclusion eligibility criteria will be listed.

#### 6.2 Demographic and Other Baseline Characteristics

#### 6.2.1 Demographics and Baseline Characteristics

The following demographics, baseline characteristics, and randomization stratification variables will be summarized by treatment group and overall.

#### Demographics:

- Sex
- Age continuous and by category  $(<65, \ge 65, <75, \ge 75, 65-74, 75-84, >85 \text{ years})$
- Ethnicity
- Race

Randomization stratification variables:





Other baseline characteristics:

Systolic and diastolic blood pressure

Other Baseline Ocular Characteristics:

- Intraocular pressure in the study eye, continuous and by category (≤21, 22-29, >29 mmHg)
- Lens status (phakic, pseudophakic, aphakic)



Ocular Imaging, OCT:

Center Subfield Thickness (CST) as evaluated by the central reading center

Ocular Imaging, Fundus fluorescein angiography (FA):

Total lesion area and CNV area

Individual-patient demographics and baseline characteristics will be listed.

## 6.2.2 Ocular and Other Medical History

Medical history includes non-ocular events and ocular events for the study and fellow (non-study) eyes. Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) [version 23.1] and will be summarized by System Organ Class (SOC) and Preferred Term (PT) for the Safety Analysis Set. Summaries will be presented by treatment group and overall. Two listings will be provided: one listing for all non-ocular medical history and an additional listing for ocular history by treatment, subject, and study/non-study eye.

#### 6.2.3 Prior and Concomitant Medications/Procedures

All medications (ocular and non-ocular) will be coded using the World Health Organization (WHO) Drug Global Dictionary, Format B3 [Version September 2020 (or a later version if updated during the study)], Anatomical Therapeutic Chemical (ATC) Classification codes. Medications will be summarized by treatment group and overall for the Safety Analysis Set. Medication summaries will be presented by Anatomical Therapeutic Chemical (ATC) class level 4 and preferred name. In addition, ocular medications will be presented separately for the study eye and fellow eye.

Prior medications and concomitant medications are defined as follows:

- Prior medications are those taken prior to the start of the first dose of study treatment
- O Concomitant medications are those with:
  - a start date on or before the last dose of study treatment and
  - a stop date after the first dose of study treatment or are ongoing at the end of the study

See Section 5.2 for imputation of missing or partial dates.

Prior and concomitant medications will be separately summarized by ocular and non-ocular for the Safety Analysis Set as follows:

- The number and percentage of patients with at least one prior / concomitant medication / procedure will be presented.
- The number and percentage of patients with at least one prior / concomitant medication / procedure within each ATC Level 4, and preferred name will be presented.
- Patients reporting use of more than one medication / procedure at each level of summarization (any medication received, ATC class, and generic drug name) will be counted only once.
- The summary will be sorted using numerical counts by descending order of Therapeutic Subgroup, then descending order of preferred name in the KSI-301 group. Where groups or terms tie will be sorted by descending order in the Aflibercept group, then alphabetically.

Prior medications and concomitant medications (ocular and non-ocular) will be listed separately for the Safety Analysis Set.

The following will be summarized and listed for concomitant medications and procedures:

- Ocular (study eye and fellow eye separately) and non-ocular concomitant medications that were initiated *before* start of treatment.
- Ocular (study eye and fellow eye separately) and non-ocular concomitant medications that were initiated *after* the start of treatment.
- Medications prescribed after study treatment discontinuation for patients who remain in the study will be listed separately.
- Concomitant ocular procedures (study eye and fellow eye separately)
   administered while patients were on study treatment will be summarized and
   listed.
- o Concomitant study eye procedures administered after study treatment discontinuation for patients who remain in the study will be listed separately.

In the listings the relative start and stop day of prior / concomitant medication (ocular and non-ocular) use will be calculated relative to the first dose date of study treatment and will be presented

for those patients who received at least one dose of treatment. If the concomitant medication is "Ongoing" it will be indicated as such in the listing and the relative stop day will not be calculated. Only original dates will be presented in the listing even though the relative day may be based on an imputed date.

#### **6.3** Protocol Deviations

All major protocol deviations will be determined and summarized by treatment group and overall. The number and percentage of patients with any major protocol deviation as well as the number and percentage of patients with deviations within each category of major deviation will be presented. The major protocol deviations will also be summarized by site. Protocol deviations will be listed in a subject data listing.

#### 7.0 EFFICACY ANALYSES

## 7.1 Primary Efficacy Analysis

#### 7.1.1 Primary Estimand

## 7.1.1.1 Target Population

The population targeted by the scientific question is treatment-naïve patients with visual impairment from wAMD.

The most relevant aspects of the study eligibility criteria for defining this population include the following key inclusion and exclusion criteria:

#### Inclusion criteria:

- 1. Active, treatment-naïve choroidal neovascularization (CNV) secondary to AMD, including subfoveal, juxtafoveal, and extrafoveal lesions, or retinal angiomatous proliferations (RAP) lesions with a CNV component that affects the central subfield, as evidenced by FA or OCT in the Study Eye at Screening.
- 2. The lesion area in the Study Eye must be <30 mm2 (12-disc areas) and can include any CNV lesion subtype.
- 3. Intra- and/or subretinal fluid and/or subretinal hyperreflective material (SHRM) affecting the central subfield of the Study Eye on OCT at Screening.
- 4. BCVA ETDRS score between 83 and 25 letters, inclusive, in the Study Eye at screening and reconfirmed at Day 1.

#### Exclusion criteria:

1. CNV secondary to other causes in the Study Eye, including pathologic myopia, angioid streaks, prior trauma, ocular histoplasmosis, or others.

- 2. Any history of macular pathology unrelated to AMD but affecting vision or contributing to subretinal or intraretinal fluid, such as central serous chorioretinopathy.
- 3. Prior treatment with any approved or investigational treatment for neovascular AMD (other than oral vitamin supplements) in the Study Eye at any time.

## 7.1.1.2 Primary Efficacy Endpoint/Variable of Interest

The primary efficacy variable of interest is BCVA, a continuous variable measured at each study visit using the ETDRS BCVA approach. The primary efficacy endpoint is the mean change in BCVA from Day 1 to the average of non-missing BCVA values of Weeks 40, 44 and 48.

## 7.1.1.3 Hypotheses and Test

The maximum clinically acceptable true difference between KSI-301 and aflibercept among wAMD patients to be considered non-inferior is 4.5 ETDRS letters, i.e. the non-inferiority margin (NI) is 4.5 letters.

The hypothesis to be tested is:

$$H_0$$
:  $\mu_K$  -  $\mu_A \le -4.5$  letters vs  $H_A$ :  $\mu_K$  -  $\mu_A > -4.5$  letters

Where  $\mu_K$  and  $\mu_A$  are the mean changes from baseline to the Weeks 40, 44 and 48 average BCVA in the KSI-301 and aflibercept groups.

If the lower limit of the two-sided 95.03% CI for the difference between the two means is >-4.5 letters, NI will be demonstrated. Furthermore, superiority will be established if the lower limit of the two-sided 95.03% confidence interval for the treatment difference (KSI-301 – aflibercept) is greater than zero.

#### 7.1.1.4 Intercurrent Events

The following intercurrent events (ICEs) may impact the assessment of the primary efficacy endpoint:

- 1. Deviations from key inclusion/exclusion criteria as defined above.
- 2. Treatment misallocation of 1 or more study treatments.
- 3. Use of prohibited medications in the study eye.
- 4. Premature discontinuation from study treatment due to study eye adverse events or due to lack of efficacy.
- 5. Premature discontinuation from study treatment due to events unrelated to study treatment such as malignancies, systemic infections, trauma, or other systemic adverse events that are not treatment-related, including discontinuations due to COVID-19.

Intercurrent events will be classified by the Sponsor prior to treatment code unmasking to prevent potential bias. Intercurrent events and the time to intercurrent events will be tabulated and listed by treatment group. Strategies for addressing the potential impact of these intercurrent events are described below.

## 7.1.2 Analysis of Primary Efficacy Endpoint

The primary efficacy endpoint will be estimated based on the FAS, i.e., all randomized subjects who received at least one treatment injection and using all available post baseline measurements or until the subject discontinues study treatment. The 'While on-Treatment' policy will be applied for the primary endpoint.

A Mixed Model for Repeated Measures (MMRM) will be used. The model assumes missing at random (MAR) and uses all available data. MMRM balances the benefits of preserving unbiased estimates because of randomization with the desire to obtain estimates for a comparison of true biological treatment effects.

The model will include the change from baseline value as the dependent variable; categorical covariates of treatment group, protocol scheduled visit, treatment × visit interaction, and the randomization stratification factors

as well as the continuous covariate of baseline BCVA value, as fixed effects; and then subject as a random effect. Within-subject correlations will be assumed to follow an unstructured covariance matrix. The change from baseline in BCVA score averaged over Weeks 40, 44 and 48 will be compared between treatment groups. The comparisons will be performed using a contrast over Weeks 40, 44 and 48.

If the model assuming an unstructured covariance matrix does not converge, a heterogeneous compound symmetry structure or an AR(1) covariance structure will be fitted.

## 7.1.3 Sensitivity Analysis 1

A sensitivity analysis, aimed at assessing the robustness of the assumptions used in the statistical model for the main estimator, will be conducted to include the FAS patients who did not have any of the following intercurrent events: deviations from key inclusion/exclusion criteria as defined above, treatment misallocations as defined above, and use of prohibited medications in the study eye during the study treatment period.

The sensitivity analysis based on this set is a type of 'Hypothetical Policy' strategy. The same MMRM as described for the primary efficacy analyses will be used.

#### 7.1.4 Sensitivity Analysis 2 (Trimmed Mean Analysis)

An additional sensitivity analysis using the trimmed mean approach (Permutt and Li 2017) will be performed.

If any of the following event types denoted by *E* occurred, patients will be considered to have the worst outcomes (defined below) and will be trimmed from the analysis:

- Discontinuation from study treatment due to study eye adverse events or due to lack of efficacy at or prior to Week 48 with no BCVA assessments available at Weeks 40, 44 and 48
- Administration of prohibited anti-VEGF medication any time during the entire treatment.

The equal trimming fraction denoted by p will be determined based on a masked assessment of the intercurrent events percentage in the study.

Patients will not be considered "to be trimmed" candidates if they have a Week 40, Week 44 and/or Week 48 assessments before the occurrence of any event type *E* above.

Patients who have no BCVA assessments available at Weeks 40, 44 and 48 due to events unrelated to study treatment such as malignancies, systemic infections, trauma, or other systemic adverse events that are not treatment-related, including discontinuations related to COVID-19 will be considered missing at random (MAR) and will be removed from the analysis.

A 95.03% confidence interval (CI) for the trimmed mean will be based on the permutation test of 30,000 generated datasets. In each dataset (random sample), the treatment assignments will be randomly permuted according to the study randomization stratification algorithm (blocked randomization stratified by

## For each generated random sample:

- An analysis of covariance (ANCOVA) model with adjustment for treatment, baseline BCVA value (continuous), as well as randomization stratification factors will be derived. The dependent variable in the ANCOVA model will be the average of non-missing values of Weeks 40, 44 and 48 BCVA change from baseline, as for the primary analysis and denoted by Y. If only one assessment is available, then the value will be used.
- 2. The value Z=Y β' X will be derived for each patient, where Y is defined above, X is the matrix for the values of the following covariates—baseline BCVA value (continuous), baseline BCVA categorical, baseline actegorical, and region; β is the ANCOVA estimated coefficient matrix for the covariates.
- 3. The Z values will be ordered and equal fractions, p, from each treatment arm will be trimmed.
- 4. The patients "to be trimmed" will always be ranked the lowest regardless of whether their adjusted values are available and trimmed from the analyses. The best (1 p)\*100 in each group will be used for the analysis specified in Step 1. If multiple patients have the same model values, they will be ranked randomly relative to each other prior to trimming.
- 5. The difference between groups in the trimmed means is derived.

Steps 1-5 are repeated 30,000 times.

The empirical permutation distribution of the difference between the trimmed means based on 2.485 and 97.515 percentiles will be derived.

If the proportion of patients "to be trimmed" in either treatment group in the permuted datasets exceeds the planned trimmed fraction p, the trimming fraction will be the maximum of the proportions of the "patients to be trimmed" in the two treatment groups.

## 7.1.5 Sensitivity Analysis 3 (Tipping Point Analysis)

A tipping point analysis will be performed where an offset (Delta based imputation penalty) is applied to the MAR imputation distribution applying a range of BCVA penalties ranging from 0.5 letter to 4.5 letters decrease (-4.5 is the non-inferiority threshold) in 0.5 letter decrements. The Delta-based multiple imputations method will pertain to the following FAS patients:

- 1. Subjects randomized to the KSI-301 arm with missing data considered missing not at random (MNAR), i.e. subjects who prematurely discontinue from study treatment due to study eye adverse events or due to lack of efficacy.
- 2. All KSI-301 treated patients with missing Week 40, 44 or 48 assessments.

The following steps will be undertaken (see Appendix 4 for the SAS syntax used and additional details).

Step 1a: A fully conditional imputation model (FCS) with predictive mean matching will be applied to all subjects' missing change from baseline BCVA values.

Step 1b: A penalty will be applied to the imputed primary efficacy endpoint for the Weeks 40, 44 and 48 in step 1a.

Fifteen complete data sets will be generated. The proposed number of imputed datasets will ensure an efficiency of at least 99% assuming a maximum of 12% rate of missing primary efficacy endpoint data using Rubin's approximation (Rubin 1987).

Step 2: a mixed model identical to the one used for the primary analysis will be run for each imputed data set.

Step 3: the mixed model mean treatment difference estimates from step 2 for all imputations are combined and Rubin's method is applied to derive an estimate of the average of Weeks 40, 44 and 48 treatment difference.

Steps 1-3 are repeated for each of the two scenario groups in the KSI-301 treatment arm and for the range of penalties in the BCVA change from baseline. The tipping point will be the penalty value that will render the lower bound of the confidence interval for mean treatment differences to be less than or equal to -4.5 letters. After the tipping point is identified, clinical judgment will determine the plausibility of the assumptions underlying this tipping point.

## 7.2 Secondary Efficacy Analyses

Table 4 lists the secondary efficacy endpoints, efficacy variable derivations, reporting statistics and analysis methods for the Final Analysis.

## 7.2.1 Analysis of Binary Data

The number and percentage of patients who gain or lose  $\geq 5$ ,  $\geq 10$  and  $\geq 15$  letters from baseline over time will be summarized by treatment group and visit, as well the number and percentage of patients with BCVA of 20/40 or better Snellen equivalent, BCVA or 20/200 or worse Snellen equivalent. The group proportions of "responders" for these categories of binary outcomes will be compared between KSI-301 and aflibercept using the Cochran–Mantel–Haenszel (CMH) test by adjusting the baseline randomization stratification factors (Section 3.3).

The number (%) of patients who fall into these categories from baseline at each post-baseline visit will be presented by treatment group, along with the weighted percentages. In addition, the weighted percentages difference between the KSI-301 and aflibercept (i.e., KSI-301 — aflibercept) and 95% CI of the difference will be presented by protocol specified visit. Percentages are calculated as 100×number of "responders"/number of patients with data at a visit. Weighted percentages are based on weighted average of observed estimates across strata using CMH weights. The CI are based on the normal approximation to the binomial proportions.

**Table 4: Secondary Efficacy Endpoints and Analysis Methods** 

| Secondary Efficacy Endpoint | Variable Derivation<br>[Source] | Summary Statistics<br>[Analysis Set] | Method of Analysis |
|---|---|---|---|
| Mean change from baseline in BCVA (ETDRS Letters) by visit over time | Continuous endpoint: Change from Day 1 to each time point [Visual Acuity Score/EDC] | LS Mean difference in change<br>from baseline at each time<br>point<br>[FAS], up to Wk 48 | Using the MMRM model (Section 7.1.2) used for deriving the primary endpoint estimate |
| Proportion of patients who gain $\geq 5, \geq 10$ and $\geq 15$ letters from baseline over time | Binary endpoints: patients had a BCVA gain ≥ 5 (yes/no); patients had a BCVA gain ≥ 10 (yes/no); patients had a BCVA gain ≥ 15 (yes/no). [Visual Acuity Score/EDC] | | |
| Proportion of patients who lose $\geq 5$ , $\geq 10$ and $\geq 15$ letters from baseline over time | Binary endpoints: patients had a BCVA loss ≥ 5 (yes/no); patients had a BCVA loss ≥ 10 (yes/no); patients had a BCVA loss ≥ 15 (yes/no). [Visual Acuity Score/EDC] | Difference in proportions (%) and 95% CI at each time point | Stratified analysis of the binary endpoint using CMH adjusting for randomization |
| Proportion of patients with<br>BCVA Snellen equivalent of<br>20/40 or better over time (≥69<br>ETDRS letters) | Binary endpoints: patients had a BCVA Snellen 20/40 or better (yes/no) [Visual Acuity Score/EDC] | [FAS], up to Wk 48 | stratification factors (Section 7.2.1) |
| Proportion of patients with BCVA Snellen equivalent of 20/200 or worse ( $\leq$ 38 ETDRS letters) over time | Binary endpoints: patients had a BCVA Snellen 20/200 or worse (yes/no) [Visual Acuity Score/EDC] | | |
| Mean change in OCT central subfield retinal thickness (CST) from baseline to the average of Weeks 40, 44 and 48 and over time | Continuous Endpoint: Change from baseline to each time point [ ] | LS Mean difference in change<br>from baseline to each time<br>point<br>[FAS], up to Wk 48 | MMRM (similar to Section 7.1.2) adjusting for baseline CST, with time, treatment, and time*treatment interaction and randomization stratification as factors Unstructured covariance matrix |

# 7.3 Exploratory Analyses

Analysis of the following exploratory endpoints may be undertaken as deemed appropriate. Intraretinal fluid (IRF) and subretinal fluid (SRF) data using AI-based grading algorithms may be explored.

**Table 5: Exploratory Efficacy Endpoints and Analysis Methods** 

| Exploratory Efficacy<br>Endpoint | Variable Derivation<br>[Source] | Summary Statistics<br>[Analysis Set] | Method of Analysis |
|---|---|---|---|
| Proportion of subjects with OCT central subfield retinal thickness (CST) < 325 microns over time | Binary endpoint: Subject with OCT CST < 325 microns (yes/no) | Difference in proportions (%) and 95% CI at each time point [FAS], up to Wk 48 | Stratified analysis of the binary endpoint using CMH adjusting for randomization stratification factors (Section 7.2.1) |
| Mean change from baseline in BCVA (ETDRS Letters) to the average of non-missing BCVA values of Weeks 40, 44 and 48 by: ≥ median vs. < median of baseline OCT-CST | Continuous endpoint: Change from baseline to average of non- missing BCVA values of Weeks 40, 44 and 48 [Visual Acuity Score/EDC] | LS Mean difference in change<br>from baseline to the average of<br>non-missing values of Weeks<br>40, 44 and 48<br>[FAS], Wks 40-48 average | Using the MMRM model (Section 7.1.2) used for deriving the primary endpoint estimate |

## 7.4 Subgroup Analyses

For each of the subgroups listed in Table 2, the primary efficacy endpoint (i.e., the change in BCVA from Day 1 to the average of Weeks 40, 44 and 48) will be analyzed using an MMRM that is described in Section 7.1.2. When a subgroup is a part of the randomization stratification variable, the corresponding stratification variable will be removed from the MMRM model as a covariate.

A forest plot will be provided to present the treatment effect of these subgroups.

#### 8.0 SAFETY EVALUATION

Safety analyses will be performed for the Safety Analysis Set. In the Final Analysis, the safety data will be summarized by treatment group.

## 8.1 Exposure to Study Medication

Study eye exposure to study medication will be summarized. Summaries will include:

- Mean (SD) and median number of injections, and number of patients receiving  $\ge 1$  injection, 1, 2, 3, 4, 5, etc. of KSI-301 or aflibercept injections.
- O Duration of study drug exposure (mean [SD] and median, in months) for subjects receiving KSI-301 5 mg or aflibercept 2 mg defined as treatment end date minus treatment start date + 1.
- o Listings will include treatment (KSI-301, aflibercept, sham) and date of injection.

A listing of patients who received study treatment other than the one assigned at randomization will include the randomized treatment, the actual administered treatment, Visit, and study Day.

#### 8.2 Adverse Events

Adverse events (AEs) will be coded to a MedDRA version 23.1 or later. AEs and Serious AEs (SAEs) will be summarized and listed by ocular events for the treated eye (or study eye), ocular events for the non-treated eye (or fellow eye), and non-ocular (systemic) events.

Adverse events with onset date on or after the initiation of study drug through the last dose date of study drug + 28 days or non-study anti-VEGF start date in study eye on or after last dose date are considered treatment-emergent AEs (TEAEs), whichever occurs first.

If the severity score of an adverse event is missing, the severity score will be imputed as severe. If the relatedness of an adverse event is missing, the adverse event will be considered related.

At each level of summarization (e.g., any AE, system organ class, and preferred term), subjects experiencing more than one TEAE will be counted only once. In the summary of TEAEs by

severity grade, subjects will be counted once at the highest severity reported at each level of summarization.

Frequency tables including patients' incidence rates will be provided for the following:

- Ocular TEAEs and treatment-emergent serious AEs (TESAEs) (study eye and fellow eye separately)
- Non-ocular TEAEs and TESAEs
- Ocular TEAEs leading to study treatment discontinuation (study eye and fellow eye separately)
- Ocular TEAEs by severity (study eye and fellow eye separately)
- o Non-ocular TEAEs by severity
- o Related ocular TEAEs (study eye and fellow eye separately) by severity
- o Related non-ocular TEAEs by severity
- Intraocular inflammation TEAEs and TESAEs not associated with infection, autoimmunity, drug toxicity, or traumatic etiologies (study and fellow eye separately)
- IOI TEAEs and TESAEs associated with infection (study and fellow eye separately)
- IOI TEAEs and TESAEs associated with autoimmune, drug toxicity, or trauma (study and fellow eye separately)
- Arteriothromboembolic (ATE) Adverse Events. ATEs will be tabulated as those events meeting the Anti-Platelet Trialists' Collaboration criteria (i.e., nonfatal myocardial infarction, nonfatal stroke, and vascular death, including deaths of unknown cause)
- o Adverse events of special interest [AESI] (study eye, fellow eye, and non-ocular separately), as defined in the protocol Section 8.3.6
- o Injection procedure related TEAEs and TESAEs (study eye)
- Non-serious TEAEs and TESAEs (study eye, fellow eye and non-ocular combined)

Adverse event data will be presented in data listings by treatment group, subject ID, and event date. Serious AEs, AEs leading to discontinuation of the study drug, intraocular inflammation events, and ATE events will be presented in separate data listings.

Adverse events from patients who remain in the study after study treatment discontinuation will be listed.

## 8.3 Deaths, Serious Adverse Events, and other Significant Adverse Events

All deaths during the study will be listed by treatment group and will include the primary cause of death. Serious AEs and other significant AEs, including those that led to interruption or withdrawal of the study drug, will be provided in separate subject data listings.

#### 8.4 Pregnancies

Listings of pregnancies, if any, and outcomes will be presented.

#### 8.5 Intraocular Pressure

For the study eye, pre- and post-injection IOP as well as the change from baseline to post baseline values will summarized, using mean, standard deviation, median, and range, by treatment group and protocol specified visit. IOP data will be listed by treatment, subject ID, study eye or non-study eye, and time point.

#### 8.6 Clinical Laboratory Evaluations

Continuous laboratory parameters will be summarized, using mean, standard deviation, median, and range by treatment group and protocol specified visit. Laboratory parameters as well as change from baseline for each parameter will be presented at Week 48.

Subjects with ALT or AST more than 3 times the Upper Limits of Normal (ULN) in combination with an elevated total bilirubin (more than 2 times the ULN); or ALT or AST more than 3 times the ULN in combination with clinical jaundice will be listed.

Other clinical laboratory results will be listed and values outside the normal ranges will be flagged along with the clinical significance.

For summary of continuous laboratory parameters, values that are lower than the LOQ will be assigned a value that is 1 unit less than the LOQ. Values that are above the LOQ will be assigned a value that is 1 unit higher than the LOQ.

#### 8.7 Vital Signs

Vital signs including pulse, systolic/diastolic blood pressure, body temperature, height, weight, and BMI will be summarized by treatment group and protocol specified visit. Descriptive statistics will be presented for results and change from baseline at each visit. Vital signs will be listed by treatment group, subject, and visit date.

#### 9.0 SAMPLE SIZE CONSIDERATIONS

The sample size for this study is based on a non-inferiority approach. The following assumptions were made in order to calculate the sample size:

- Overall Type I error rate of 0.025. Testing at the 0.025 level for non-inferiority corresponds to setting 95% CIs.
- Statistical power of >90%.
- Standard deviation of the distribution of change in visual acuity from baseline of letters.
- Actual expected mean treatment difference between treatments of at most -0.3 letters
- The maximum clinically acceptable true difference for KSI-301 to be considered non-inferior, or the "non-inferiority margin", is 4.5 letters.
- The statistical test used to compare the two treatment arms is an independent t-test on the mean change in visual acuity from baseline.
- Lost to follow-up/dropout rate of approximately

The sample size calculated using the above assumptions is approximately 500 patients (250 per treatment arm).

# 10.0 SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

No changes in the conduct of the study have occurred relative to the latest version of the protocol at this time.

In this SAP, the Sponsor has defined the primary estimand, analysis populations, and strategies for addressing intercurrent events, missing data, and a set of sensitivity analyses for the primary efficacy outcome. Where relevant, these definitions take precedence over those defined in the study protocol.

Also in this SAP, the Sponsor has clarified that the non-inferiority margin will be 4.5 letters for the primary efficacy endpoint and corresponding sensitivity analyses per the FDA's draft guidance on wAMD drug development dated February 2023.

#### 11.0 REFERENCES

US Food and Drug Administration Guidance Document - E9(R1) Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials (May 2021). Available at https://www.fda.gov/media/148473/download.

US Food and Drug Administration Guidance Document – Non-Inferiority Clinical Trials to Establish Effectiveness (November 2016). Available at <a href="https://www.fda.gov/media/78504/download">https://www.fda.gov/media/78504/download</a>.

US Food and Drug Administration Draft Guidance Document – Neovascular Age-Related Macular Degeneration: Developing Drugs for Treatment (February 2023). Available at <a href="https://www.fda.gov/media/165606/download">https://www.fda.gov/media/165606/download</a>.

Rubin, D.B. (1987) Multiple Imputation for Nonresponse in Surveys, New York, John Wiley and Sons.

Littell, Ramon C., George Milliken, Walter W. Stroup, Russell D. Wolfinger, and Oliver Schabenberger (2006) SAS<sup>(R)</sup> for Mixed Models, 2<sup>nd</sup> Edition (2006), SAS Institute, Cary NC.

Little, R.J.A. and Rubin, D.B. (2002). Statistical Analysis with Missing Data, 2<sup>nd</sup> edition, New York: John Wiley.

SAS/STAT® 14.1 User's Guide The MIANALYZE Procedure, SAS institute, Cary, NC, available online at https://support.sas.com/documentation/onlinedoc/stat/141/mianalyze.pdf

SAS/STAT® 14.1 User's Guide The MI Procedure, SAS institute, Cary, NC, available online at https://support.sas.com/documentation/onlinedoc/stat/141/mi.pdf.

van Buuren, Stef Flexible Imputation of Missing Data, 2nd Edition (2018).

Permutt T, Li F. Trimmed means for symptom trials with dropouts. Pharm Stat. 2017

#### 12.0 APPENDICES

Appendix 1: Schedule of Activities

# **Appendix 1: Schedule of Activities**

| Visit | Screening | Day<br>1 | Week<br>2 | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 | Week<br>28 | Week<br>32 | Week<br>36 | Week<br>40 | Week<br>44 | Week<br>48/ET | Week 52 <sup>13</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Windows (days) | D-21 to<br>D-1 | | +/-3 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 |
| Informed consent | X | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | |
| Medical & Ocular History | X | | | | | | | | | | | | | | | |
| Inclusion/Exclusion Criteria | X | X | | | | | | | | | | | | | | |
| Concomitant Medication<br>Review <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| AE/SAE Review <sup>2</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| General Assessments | | | | | | | | | | | | | | | | |
| Vital signs <sup>3</sup> | X | X | | | | | | | | | | | | | X | |
| Laboratory <sup>4</sup> | X | | | | | | | | | | | | | | X | |
| Plasma ADA samples <sup>5</sup> | | X | | X | | | | X | | | | | | | X | |
| Plasma PK/biomarker<br>samples <sup>5</sup> | | X | X | X | | | | X | | | | | | | X | |
| Pregnancy test <sup>6</sup> (WOCBP only) | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Ophthalmic Assessments <sup>7</sup> | | | | | | | | | | | | | | | | |
| BCVA ETDRS (4 meters) <sup>8</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| | | X | | | | | X | | | | | | | | | |

| Visit | Screening | Day<br>1 | Week<br>2 | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 | Week<br>28 | Week<br>32 | Week<br>36 | Week<br>40 | Week<br>44 | Week<br>48/ET | Week 52 <sup>13</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Windows (days) | D-21 to<br>D-1 | | +/-3 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 | +/-7 |
| Ophthalmic exam (Slit-<br>lamp, IOP <sup>9</sup> , dilated indirect<br>ophthalmoscopy) | х | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| SD-OCT <sup>10</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Color Fundus photos <sup>10</sup> | X | | | | | | | | | | | | | | X | |
| Fluorescein angiogram <sup>10</sup> | X | | | | | | | | | | | | | | X | |
| Randomized study treatment<br>(KSI-301, aflibercept or<br>sham) per IRT designation <sup>11</sup> | | X | | X | X | X | X | X | X | X | X | Х | X | X | | |
| Post-injection Assessments<br>(vision check, IOP <sup>9</sup> ) <sup>12</sup> | | X | | X | X | X | X | X | X | X | X | X | X | X | | |

- Abbreviations: ADA = anti-drug antibody; AE = adverse event; BCVA = best corrected visual acuity; ET = early termination; ETDRS = early treatment diabetic retinopathy study; IRT = interactive response technology; PK = pharmacokinetics; SAE = serious adverse event; SD-OCT = spectral domain optical coherence tomography; WOCBP = women of childbearing potential.
- Record any concomitant medication used by the participant within 30 days prior to Day 1. Procedural medications administered (e.g., dilating drops, fluorescein) will not be recorded.
- After informed consent has been obtained but prior to initiation of study intervention, only serious adverse events caused by a protocol-mandated intervention should be reported. After initiation of study intervention (Day 1), all AEs will be reported until the final study visit or the ET visit if applicable. See protocol Section 8.3.1.
- <sup>3</sup> Height and weight are taken at screening only.
- <sup>4</sup> Clinical laboratory test as described in Appendix 2 and Table 4.
- <sup>5</sup> Blood draws for ADA, plasma PK, and biomarker samples are to be taken pre-injection.
- Urine pregnancy test will be performed locally for women of childbearing potential, prior to fluorescein angiogram and study treatment (if applicable). If urine pregnancy test is positive, it must be confirmed with a serum pregnancy test. Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/IEC.
- Ophthalmic assessments will be performed in both eyes at Screening and Week 48, and in the Study Eye only at all other timepoints.
- <sup>8</sup> Perform BCVA before any other ophthalmic assessments and prior to dilation.
- <sup>9</sup> Method used to measure IOP must remain consistent throughout study.
- 10 It is mandatory that the same model of device is used for the entire duration of the study.
- Participants who discontinue study treatment should NOT be considered withdrawn from the study. Additional details are provided in protocol Section 7.1.
- Post injection assessments include vision check for counting fingers and tonometry. The post-injection assessments should be performed by unmasked assessors.
- Week 52 is a final safety assessment that will be done via telephone call for all participants, except in WOCBP, in which case a site visit is required for the safety assessment that includes a pregnancy test.









